CLINICAL TRIAL: NCT05933681
Title: Neurophysiology Biomarkers of Cognitive Impairment Associated With Deep Brain Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sarah Bick, Assistant Professor of Neurosurgery, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 230539
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Parkinson Disease; Cognitive impairment; Movement Disorders; Brain Diseases
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Movement Disorders; Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Determination of DLPFC neurophysiology biomarkers of DBS associated cognitive impairment (Experimental): Neurophysiology recordings will be performed from dorsolateral prefrontal cortex (DLPFC) during deep brain stimulation surgery, with and without STN or GPI stimulation, at rest and during a working memory task.
  Interventions: Device: Neural recordings and stimulation
- Neurophysiology biomarkers of DBS mediated cognitive impairment following chronic stimulation (Experimental): Neurophysiology recordings will be performed from subthalamic nucleus (STN) or globus pallidus internus (GPI) with stimulation on and off, at rest and during a working memory task, in patients who have previously been implanted with DBS and have implantable pulse generators capable of recording local field potentials.
  Interventions: Device: Neural recordings and stimulation

INTERVENTIONS:
Device: Neural recordings and stimulation — Neural activities from the dorsolateral prefrontal cortex and implanted DBS generator will be recorded, during resting and working memory tasks, and with the DBS target turned on and off.

SUMMARY:
The study aims to investigate cognitive impairment associated with Deep Brain Stimulation (DBS) in Parkinson's Disease patients, with a focus on identifying neurophysiology biomarkers of DBS associated cognitive changes. Using neurophysiology data recorded during DBS surgeries and post-implantation, the research intends to identify biomarkers in order to optimize electrode placement, enhance programming, and ultimately minimize DBS-related cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

• Scheduled to undergo deep brain stimulation surgery under local anesthesia at Vanderbilt University Medical Center (Arm 1)

* Active deep brain stimulation system with implantable pulse generator capable of recording local field potentials (Arm 2)
* Diagnosis of Parkinson's disease as determined by a movement disorders specialist neurologist
* Age at least 18
* Able to participate in intraoperative testing
* English speaking

Exclusion Criteria:

* Age less than 18
* Not able to participate in intraoperative testing (ex unable to comprehend instructions or follow directions)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Determination of DLPFC beta power a biomarker of DBS associated cognitive impairment in the acute stimulation setting | Baseline to end of Deep Brain Stimulation (DBS), approximately 3-4 hours
  Working memory tasked will be conducted during surgery, and local field potentials (LFPs) will be recorded from the DLPFC both at rest and during task execution, under two conditions: with and without stimulation.
Determination of STN local field potential biomarkers of DBS mediated cognitive impairment following chronic stimulation | 1 hour
  Local field potentials will be recorded from subthalamic nucleus or globus pallidus internus in patients with an existing DBS system with implantable pulse generator capable of recording local field potentials. Recordings will be performed at rest and during a working memory task, with DBS on and off.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Bick, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No